CLINICAL TRIAL: NCT04525170
Title: Clinical Evaluation of Hydra-PEG (Polyethylene Glycol) Treatment (HPT) Treated Rigid Contact Lenses Made From Hexafocon A
Brief Title: Clinical Evaluation of HPT Treated Rigid Contact Lenses Made From Hexafocon A
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: It was decided by the sponsor to not proceed.
Sponsor: Contamac Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CM-002-002
Record Dates: First submitted 2015-10-02; First posted 2020-08-25 (Actual); Last update posted 2020-08-25 (Actual); Status verified 2020-08

CONDITIONS: Ametropia
MeSH Terms: conditions — Refractive Errors | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HPT treated (Experimental): daily wear Hexafocon A rigid contact lens treated with Hydra PEG surface coating
  Interventions: Device: HPT treatment
- untreated (Experimental): daily wear Hexafocon A rigid contact lens
  Interventions: Device: untreated

INTERVENTIONS:
Device: HPT treatment
  Other Names: Hydra-PEG (Polyethylene Glycol) Treatment
  Arms: HPT treated
Device: untreated
  Arms: untreated

SUMMARY:
This will be an up to six months, subject-masked, contralateral, parallel-group, randomised, daily wear study. All subjects will wear the Test lens in one eye and the Control lens in the other eye. Data from the first four weeks of Test and Control lens exposure will be used for the FDA 510 (k) submission.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to sign the informed consent form
* Aged ≥18 years old
* Experienced wearer of rigid gas permeable contact lenses
* Subject's habitual contact lenses must be made of Boston XO (hexafocon A) material
* Subjects must have owned spectacles or contact lenses prior to enrolment for this trial
* Spherical power between -10.00 D and +10.00 D (at vertex distance 0 mm)
* Corneal astigmatism ≤2.00 D

Exclusion Criteria:

* Eye injury or surgery within 3 months immediately prior to enrolment for this trial
* Pre-existing ocular irritation that would preclude contact lens fitting
* Currently enrolled in an ophthalmic clinical trial
* Evidence of systemic or ocular abnormality, infection or disease which is likely to affect successful wear of contact lenses or use of the accessory solutions, as determined by the investigator
* Any use of medications for which contact lens wear could be contradicted, as determined by the investigator
* Current extended-wear users (sleep-in overnight)
* Current monovision lens wearers
* Current wearers of multifocal contact lenses
* Current wearers of toric contact lenses (front surface design)
* Current wearers of astigmatic contact lenses (posterior surface design)
* Has a reported "Strong" comfort or vision preference between each eye with their habitual RGP lenses
* Unacceptable fit of habitual lenses
* Pregnant women and nursing mothers
* Best-corrected visual acuity worse than 6/9 (LogMAR: +0.20; Snellen decimal: 0.63)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
questionnaire addressing subjective comfort and wear time | subjects will be followed-up for one month
  Subjects rated on a scale from 1 to 10, where 1 was 'poor' and 10 was 'excellent'.
limbal redness - ocular biomicroscopy | subjects will be followed-up for one month
  Findings were graded based on a grading scale which ranged from 0 to 4, where 0 is none, 1 is trace, 2 is mild, 3 is moderate and 4 is severe.
corneal staining - ocular biomicroscopy | subjects will be followed-up for one month
  Findings were graded based on a grading scale which ranged from 0 to 4, where 0 is none, 1 is trace, 2 is mild, 3 is moderate and 4 is severe.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Hartwig, PhD, Principal Investigator — Hartwig Research Center
Locations (2):
- Germany (2):
  - Hartwig Research Center, Heikendorf, S-H
  - Siehste, Kassel